CLINICAL TRIAL: NCT03794557
Title: A Phase 2, Single-Center, Double-Blind, Placebo-Controlled, Study of PUL-042 Inhalation Solution in Rhinovirus-induced Symptoms in Current Smokers With Gold Stage 0 Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: The Effect of Inhaled PUL-042 on Rhinovirus-induced Symptoms in Smokers With GOLD Stage 0 COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pulmotect, Inc. (Industry)
Collaborators: Imperial College Healthcare NHS Trust (Other); VirTus Respiratory Research Ltd (Unknown); MWB Consulting Ltd (Unknown); Data Magik Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PUL-042-402
Record Dates: First submitted 2018-12-24; First posted 2019-01-07 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PUL-042 (Experimental): PUL-042 Inhalation Solution
  Interventions: Drug: PUL-042 Inhalation Solution
- Placebo (Placebo Comparator): Sterile Water for injection
  Interventions: Drug: Sterile Water Injection

INTERVENTIONS:
Drug: Sterile Water Injection — Inhaled Sterile Water Injection
  Arms: Placebo
Drug: PUL-042 Inhalation Solution — PUL-042 Inhalation Solution
  Arms: PUL-042

SUMMARY:
This is a study examining the effect of inhaled PUL-042 on peak lower respiratory symptoms as measured by subject diary in early stage COPD subjects who are experimentally infected with rhinovirus.

Subjects will receive 1 dose of PUL-042 followed by inoculation with HRV A16 virus 24 hours later. An additional dose of PUL-042 will be administered 48 hours post-inoculation. Subjects will be followed for 6 weeks post-inoculation

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled Phase 2 study examining the effects of inhaled PUL-042 on Lower Respiratory Symptom Score (LRSS) in GOLD stage 0 COPD patients.

Smoking subjects (>10 pyh) with symptoms suggestive of early COPD (cough, sputum production but normal spirometry, meeting GOLD 0 criteria) will be screened. Following screening (days -21 to -11 prior to infection), eligible subjects will be enrolled and will undergo a baseline sampling visit on study day -8 and will complete questionnaires from study day -8 to -2 (7 days total) recording their baseline symptoms

There will be two treatment arms in the study. The arms will be:

* Placebo administered on study day -1 and study day 2
* PUL-042 administered on study day -1 and PUL-042 administered on study day 2

On day 0 subjects will be experimentally infected with HRV A16 (100 TCID50) via an atomizer to the upper airway. Subjects will subsequently be required to attend the clinic on study days 1-7, 9, 12, 15, 21 and 42 for follow up visits. Subjects will continue their diaries at home during the period when not attending clinic visits, namely days 8, 10, 11, 13, 14, 16-20 and 22-41.

Spirometry assessments will be conducted by clinic staff on clinic visit days. PEF, FEV1, FVC and FEV1/FVC ratio will be completed at the visit using the clinic study-supplied spirometry equipment.

Sputum samples and serum will be analyzed for inflammatory markers. Serum samples will be obtained from subjects at screening and during clinic visits on study days -1, 0, 2, 3, 5, 7, 9, 12, 15, 21 and 42. Sputum samples will be obtained at baseline (BL) and on study days -1, 0, 2, 5, 7, 9, 12, 15, and 21.

Nasal lavage samples will be collected during baseline (BL) and on study days -1, 0, 1-7, 9, 12, 15, 21 and 42 for assessment of virus load and pro-inflammatory cytokines etc. in the upper airway.

Subjects will be asked to complete the following questionnaires on days -8 to day 42 during the study:

1. The lower respiratory symptom scores as measured by Mallia
2. The upper respiratory symptoms measured by the Jackson score as measured by Mallia
3. The COPD Assessment Test (CAT) score
4. The EXACT-RS Lower Respiratory Symptom questionnaire
5. The Wisconsin Upper Respiratory Symptom Survey-11 (WURSS-11)
6. Subjects will record any medication use in a specific diary.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, with symptoms (cough, sputum production) suggestive of GOLD stage 0 COPD for at least one year prior to the screening visit in accordance with the GOLD 2014 guidelines;
* Current smokers with >10 pyh;
* Subject has risk of COPD defined by GOLD Staging Criteria level 0 where the subjects' post-bronchodilator FEV1/FVC ratio >0.70 and FEV1 is >80% normal predicted;
* CAT score at screening >3 and < 15;
* Sero-negativity to HRV A16 neutralizing antibody;
* Patients together with their partners of reproduction potential (males and females) must practice an acceptable method of birth control with a failure rate of a Pearl index of less than 1% per year, to be used consistently and correctly throughout the course of the study.
* Ability to understand and give informed consent.

Exclusion Criteria:

* Sero-positivity to HRV A16
* Use of systemic or nasal topical steroids, inhaled corticosteroids (ICS), systemic immunosuppressants, antibiotics, LABA, and LAMA and oral theophylline and/or roflumilast within 30 days;
* Subjects with evidence of an upper or lower respiratory infection within 6 weeks;
* A history or current evidence of bronchiectasis, cystic fibrosis, interstitial lung disease or other significant chronic lung disease;
* A history within the last 5 years or current evidence of carcinoma of the bronchus;
* A history within the last 5 years or current evidence of asthma;
* A history of active tuberculosis or history of significant lung disease as a result of previous tuberculosis infection;
* A medical history or current clinical evidence of significant hematological, gastrointestinal, renal, hepatic, cerebrovascular, immunologic, psychiatric or cardiovascular disease or event (including uncontrolled hypertension as determined by the Investigator), or any clinical condition that may, in the opinion of the Investigator or Medical Monitor, impact on the subject's ability to participate in the study;
* Clinical laboratory values at screening for neutrophils, hemoglobin and hematocrit which reflect grade 2 or higher reductions from normal range, or ALT results which reflect grade 2 or higher elevations per the 'CTCAE' guidelines. Subjects with other clinical laboratory abnormalities outside normal reference ranges will be considered for inclusion, if in the opinion of the Principal Investigator or Medical Monitor the abnormalities are not clinically significant, or will not jeopardize the safety of the subject or the validity of the study;
* Use of cold preparations, anti-cholinergics, nasal lavage preparations or sprays, cough medications, or prescription or over-the-counter nasal decongestants within 30 days;
* Current abuse of alcohol or illicit drugs, or history of alcohol or illicit drug abuse within the preceding 2 years;
* A positive pregnancy test at screen;
* Received an investigational drug or vaccine within 30 days or 5 half-lives (whichever is longer), or use of an investigational medical device within 30 days prior to the screening visit or in the interval between screening and study day -1;
* Inability to tolerate nebulization based on the Principal Investigator's medical judgment or a ≥12% drop in FEV1, at either 15 or 30 minutes after the completion of administration of a dose of nebulization test solution (SWFI) of the same volume and under the same nebulization conditions that is planned to be used for study drug administration, compared to the FEV1 obtained immediately prior to administration of the nebulization test solution.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Lower Respiratory Symptom Score as measured by Mallia et al (Am J Respir Crit Care Med. 2011) | Daily Scores Day 0-42
  The peak daily lower respiratory symptom score as measured by Mallia recorded in the 6 weeks post-infection period. This is a measure of a number of lower respiratory symptoms in a 24 hour period that include: shortness of breath (scale 0-4; 0 = not breathless, 4 = breathless at rest) wheeze (0-4; 0 = no wheeze, 4 = wheeze at rest), cough (0-3; 0 = no cough, 3 = severe cough), sputum quantity (0-3; 0 = none, 3 = large volume , more than 100 ml) sputum quality (0-3; 0 = none, 3 = purulent, green in colour). The total lower respiratory symptom score is the sum of all the above measurements (minimum 0, maximum 17) recorded on each day. These values will be recorded via a study diary over a six week period (day 0-42). Peak value is the highest daily total value over the 6 week post-infection period.

SECONDARY OUTCOMES:
Lower Respiratory Symptoms | Daily Scores Days 0-42
  The EXAcerbations of Chronic obstructive disease Tool-Respiratory Symptoms (EXACT-RS)
Lower Respiratory Symptoms | Daily Scores Days 0-42
  COPD Assessment Test (CAT)
Upper Respiratory Symptoms | Daily Scores Days 0-42
  Jackson Score as measured by Mallia et al (Am J Respir Crit Care Med. 2011). A modified Jackson score will be utilized which assesses the following eight upper respiratory symptoms daily: nasal congestion, runny nose, sneezing, cough, sore throat, general malaise, headache, chilliness (each scored 0-3 where 0 = none, 3 = severe). Minimum daily score= 0, maximum daily score= 24.
Upper Respiratory Symptoms | Daily Scores Days 0-42
  Wisconsin Upper Respiratory Symptom Survey-11 (WURSS-11)
Lung Function | Days 0-42
  Peak Expiratory Flow (PEF) L/min
Lung Function | Days 0-42
  Forced Expiratory Volume in 1 Second (FEV1) L/second
Lung Function | Days 0-42
  Forced Vital Capacity (FVC) L
Lung Function | Days 0-42
  FEV1/FVC ratio
Inflammatory Mediator | Days 0-42
  CXCL 10/IP-10 measured by ELISA in nasal secretions, sputum and serum. Results reported in pg/mL
Inflammatory Mediator | Days 0-42
  IL-6 measured by ELISA in nasal secretions, sputum and serum. Results reported in pg/mL
Number of successfully infected patients | Days 0-42
  Detectable virus load; seroconversion

CONTACTS AND LOCATIONS:
Overall Officials: Onn Min Kon, MD, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust, St Mary Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mallia P, Message SD, Gielen V, Contoli M, Gray K, Kebadze T, Aniscenko J, Laza-Stanca V, Edwards MR, Slater L, Papi A, Stanciu LA, Kon OM, Johnson M, Johnston SL. Experimental rhinovirus infection as a human model of chronic obstructive pulmonary disease exacerbation. Am J Respir Crit Care Med. 2011 Mar 15;183(6):734-42. doi: 10.1164/rccm.201006-0833OC. Epub 2010 Oct 1. PMID 20889904